CLINICAL TRIAL: NCT04285177
Title: Effect of Strabismus Surgery on Macular and Subfoveal Choroidal Thickness Assessed by Spectral Domain Optical Coherence Tomography
Brief Title: Choroidal and Retinal Thickness Following Strabismus Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Heba Shafik, Clinical Associate Professor, Tanta University
Other Study IDs: TUORU003
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Strabismus; Retinal Thickening
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Horizontal muscle surgery: Patients suffering from esotropia or exotropia, will have medial/lateral rectus recession/resection
  Interventions: Procedure: Strabismus surgery
- Patients with Inferior Oblique Overaction: Will undergo inferior Oblique Myectomy
  Interventions: Procedure: Strabismus surgery
- Patients with combined horizontal and oblique muscle surgery: Having combined surgery
  Interventions: Procedure: Strabismus surgery

INTERVENTIONS:
Procedure: Strabismus surgery — Resection or recession of the medial or lateral rectus muscle, or inferior oblique myectomy

SUMMARY:
Prospective study, conducted at Tanta University Ophthalmology Department Measurement of macular and choroidal thickness before and after strabismus surgery

DETAILED DESCRIPTION:
This is a prospective study and will be conducted in Tanta University hospital

* Duration: February 2020 till May 2020 and may be extended
* The study will include 30 patients who suffer from esotropia or exotropia, inferior oblique (IO) over-action with or without any other type of horizontal deviation

Pre-operative measurement of the macular and choroidal thickness by Enhanced Depth Imaging Optical Coherence Tomography (EDI-OCT).

Post-operative measurement: First day, first week, one month then 3 months.

ELIGIBILITY:
Inclusion Criteria:

* No prior history of ocular surgery or trauma
* Normal ocular examination findings
* No medical or family history of retinal disease, glaucoma or diabetes mellitus.

Exclusion Criteria:

* Patients with orbital and/or craniofacial abnormalities
* Patients with sensory or restrictive strabismus or neurological disease
* Preoperative retinal or macular pathology
* Patient who is unable to cooperate to do OCT scanning

Ages: 7 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All individual with strabismus fulfilling the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Choroidal and retinal thickness change after strabismus surgery | preoperative, 1st week, 1st month, and 3 months
  Measured by Spectral Domain Optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Sharif Y El Emam, MD, Principal Investigator — Tanta University
Locations (1):
- Tanta University Hospital, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No